CLINICAL TRIAL: NCT01553253
Title: From Acute To Chronic Postoperative Pain in Patients for Elective Cholecystectomy: The Significance of Components of Pain
Brief Title: From ACute To Chronic Postoperative Pain in Patients for Elective Cholecystectomy
Acronym: FACTS1
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Region of Southern Denmark (Other); Vejle Hospital (Other); Manufacturer Mads Clausen Foundation (Other); DASAIMS Forskningsinitiativ (Unknown); Fonden Else Poulsens Mindelegat (Unknown); Oberstinde Kirsten Jensa la Cours Foundation (Other); Læge Frk. K. Rasmussens Mindelegat (Unknown)
Responsible Party: Principal Investigator, Morten Rune Eckhardt, Afdelingslæge, Ph.D.-student, Odense University Hospital
Other Study IDs: FACTS1
Record Dates: First submitted 2012-03-02; First posted 2012-03-14 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Postcholecystectomy Pain; Chronic Postoperative Pain; Visceral Pain; Referred pain; Somatic pain; Quantitative Sensory Testing
MeSH Terms: conditions — Pain; Pain, Postoperative; Visceral Pain; Pain, Referred; Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic Pain is a wellknown complication after cholecystectomy. Intensity of the pain in the first week after the operation is a predictive factor for the development of chronic pain, but it is unknown whether the risk is more related to one of the different components of acute pain (ie somatic, visceral, referred). Furthermore the chronic pain has not been systematically described in terms of type of pain or sensory abnormalities etc. (allodynia, hyperalgesia etc.).

The purpose of the study is to examine whether intensity of components of acute pain is predictive for development of chronic pain after cholecystectomy and to characterize the chronic pain by quantitative sensory testing.

DNA-samples are collected to examine genetical factors, important for perception of pain, and the development of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective cholecystectomy
* 18 years or older at the day of the operation
* Capable of speaking, reading and writing danish

Exclusion Criteria:

* Previous abdominal operation
* Patients with preoperative neuropathies
* Patients with other diseases in the nervous system, preoperative paresthesias or other sensory disturbances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive Patients for elective cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | 12 months

SECONDARY OUTCOMES:
Quantitative sensory testing values in referred pain area. | 12 Months
  Quantitative sensory testing values in referred pain area compared to contralateral side and preoperative values.
  The following quantitative sensory tests are performed:
  Cold Detection Threshold,Warm Detection Threshold, Cold Pain Threshold, Heat Pain Threshold, Mechanical detection Threshold, Mechanical Pain Threshold, Allodynia, Hyperalgesia, Wind-Up Ratio, Vibration Detection Threshold, Pressure Pain Threshold
Abdominal pain | 6 months
Quantitative sensory testing values in referred pain area. | 6 Months
  Quantitative sensory testing values in referred pain area compared to contralateral side and preoperative values.
  The following quantitative sensory tests are performed:
  Cold Detection Threshold,Warm Detection Threshold, Cold Pain Threshold, Heat Pain Threshold, Mechanical detection Threshold, Mechanical Pain Threshold, Allodynia, Hyperalgesia, Wind-Up Ratio, Vibration Detection Threshold, Pressure Pain Threshold

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Odense University Hospital, Nyborg
  - Lillebælt Hospital, Vejle